CLINICAL TRIAL: NCT02102165
Title: AURORA: Aiming to Understand the Molecular Aberrations in Metastatic Breast Cancer.
Acronym: AURORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Breast International Group (Other)
Collaborators: Jules Bordet Institute (Other); Frontier Science & Technology Research Foundation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BIG 14-01; 1408-BCG (Other: EORTC); GBG 85 (Other: German Breast Cancer Group (GBG)); ICR-CTSU/2014/10050 (Other: The Institute of Cancer Research, UK)
Record Dates: First submitted 2014-03-19; First posted 2014-04-02 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer
Keywords: Aurora; breast cancer; metastatic; molecular screening; targeted gene sequencing; molecular aberrations; exploratory; biomarker
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- metastatic lesion biopsy (Experimental): biopsy of metastatic lesion will be performed at program inclusion or maximum 6 months prior to inclusion. Sample of primary tumor must be available at inclusion.
  Interventions: Procedure: metastatic lesion biopsy

INTERVENTIONS:
Procedure: metastatic lesion biopsy — a medical test commonly performed by a surgeon or an interventional radiologist in order to collect tissues for examination; in this case from a metastatic lesion

SUMMARY:
This program initially aims to recruit 1300 breast cancer patients from a large number of hospitals across Europe. Eligible patients are those who are 18 or older, either female or male, and who have not received more than 1 type of treatment from the time metastases were discovered, metastasi(e)s has just been diagnosed or their disease has come back (disease relapse). Biopsy samples from both the primary and metastatic (or relapsed) tumor will be collected for central analyses, together with blood, serum and plasma samples. Any samples not analyzed immediately will be stored in an independent bio-repository to enable future (not yet defined) research aimed at better understanding metastatic breast cancer.

In summary, the main objectives of AURORA are to better understand the genetic aberrations in metastatic breast cancer and to discover the mechanisms of response or resistance to therapy, in order to ultimately identify the "right therapy for each individual patient". At the same time, patients with genetic aberrations that are being targeted by new drugs in development will be offered the possibility to participate in clinical trials, when approved and available in their countries. Ultimately, the aim of AURORA is to improve the outcomes of all patients diagnosed with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male ≥ 18 years with diagnosis of locally recurrent/advanced BC not amenable to treatment with curative intent or MBC who have not received more than 1 line of systemic therapy (any type) in the metastatic setting.

   Under protocol 4.0, eligible patients will be limited to locally recurrent/advanced breast cancer not amenable to treatment with curative intent or MBC with:
   * histopathology-confirmed TNBC as defined by ER <1% and HER2 negative following ASCO-CAP guidelines
   * ILC (either based on ILC morphology or negative E-cadherin expression confirmed by IHC). Mixed ILC/invasive ductal carcinoma are not eligible for the ILC cohort.
   * late relapse BC (any subtype). Late relapse is defined as a patient with a radiologic or histologic confirmation of advanced or MBC relapse > 10 years from the primary BC diagnosis.
2. Written informed consent prior to registration into the program.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
4. Availability of primary tumor tissue for research purposes.
5. Patient must have a metastatic lesion accessible for biopsy and must agree with the biopsy procedure.

   1. Up until protocol 3.0, up to 100 patients with bone-only metastasis have been included without a metastatic biopsy, if plasma samples have been collected at screening, and if the patient met all other eligibility criteria.
   2. In protocol 4.0, metastatic tumor biopsies from bone lesions will be accepted provided that the chosen site of biopsy was not previously irradiated.
   3. Brain tissue is accepted if it is obtained through surgical excision not planned for AURORA, but as part of the routine clinical practice.
6. The biopsy of the metastatic lesion must be conducted either at the initial diagnosis of the BC relapse before the initiation of 1st line systemic therapy or at the 1st disease progression before initiation of a second line systemic treatment. There is no restriction in the type of therapeutic modality considered as 1st line systemic treatment, which can consist of any type of treatment administered after the diagnosis of the advanced BC relapse till the 1st disease progression thereafter.
7. Biopsies obtained during routine clinical practice are accepted if both formalin-fixed paraffin-embedded (FFPE) and Frozen Tissue (FT) blocks were collected concurrently from the same metastatic lesion and if collected at the pre-specified timelines for AURORA.
8. Availability of a whole blood, serum and plasma samples collected at the time of screening.
9. Patient agrees to provide blood samples at regular intervals, from the screening as well as during the follow-up phase of the program.

Exclusion Criteria:

1. The patient has received more than 1 line of systemic therapy (any type) in the metastatic setting.
2. Patients who have received prior palliative radiotherapy to the only site that is accessible to biopsy.
3. Presence of severe hematopoietic, renal, and/or hepatic dysfunction, including but not restricted to albumin < 3 g/dl.
4. Known increased risk of hemorrhage during biopsy procedure, as evaluated by the treating physician.
5. Previous or current malignancies of other histologies within the last 5 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Metastatic Breast Cancer (MBC) understanding | 1 year after end of acrrual
  To improve the understanding of locally recurrent/advanced BC and MBC by using high-throughput technologies on primary, metastatic, as well as plasma ctDNA samples, to explore tumor heterogeneity, clonal evolution and transcriptional changes associated with mutational and copy number variation (CNV) patterns.

SECONDARY OUTCOMES:
Identification of "exceptional responders" and "rapid progressors"; the outlier patients | 1 year after end of accrual and subsequently during follow up period of 10 years
  To discover biomarkers of response and/or resistance to systemic therapy using genomic and transcriptomic data of "exceptional responders" and "rapid progressors" (collectively referred to as "outliers", as defined in the AURORA protocol).
Feasibility of implementing a global molecular screening platform for MBC | 1 year after end of accrual
  To provide evidence that can contribute in assessing the feasibility of implementing a global molecular screening platform of MBC
Patient identification to match with biomarker-driven clinical trials | on ongoing basis during 3 years' patient recruitment
  To identify patients with candidate driver alterations in their tumors that can be matched to biomarker-driven clinical trials.
Building new therapeutic hypotheses | 1 year after end of accrual and subsequently during follow up period of 10 years
  To build new therapeutic hypotheses based on findings generated by Targeted Gene Sequencing (TGS).
Patients' prognosis determination | 1 year after end of accrual and subsequently during follow up period of 10 years
  To evaluate the prognostic relevance of genomic alterations detected in plasma ctDNA samples, tumor metastatic biopsies and archived primary tissue.
Correlation between molecular alterations and standardly assessed efficacy endpoints | 1 year after end of accrual and subsequently during follow up period of 10 years
  To correlate molecular alterations in patients with the efficacy endpoints (response rate, progression-free survival and overall survival).

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Aftimos, MD, Principal Investigator — Institut Jules Bordet, Brussels, Belgium; Angel Guerrero Zotano, MD, Principal Investigator — Instituto Valenciano de Oncologia, Valencia, Spain; Matteo Benelli, PhD, Principal Investigator — Breast International Group
Locations (52):
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - Grand Hopital Charleroi, Charleroi
  - UZ Leuven, Leuven
  - CHU de Liège, Liège
  - Clinique et Maternité Sainte-Elisabeth (CMSE - Namur), Namur
- Germany (2):
  - Kliniken Essen-Mitte, Klinik für Senologie/ Brustzentrum, Essen
  - Frauenkliniken Maistrasse-Innenstadt und Großhadern, München
- Landspitali, Reykjavik, Iceland
- Italy (9):
  - Ospedale degli Infermi - S.O.C.Oncologia, Biella
  - Ospedale di Bolzano - Oncologia Medica, Bolzano
  - Ospedale Ramazzini di Carpi, Carpi
  - IRCCS AOU San Martino-IST, Genova
  - ULSS 21 Legnago, Legnago
  - Istituto Europeo di Oncologia, Milan
  - UOC Oncologia Medica - AOU Parma, Parma
  - Fondazione Salvatore Maugeri, Pavia
  - IRCCS Az Ospedaliera S.Maria Nuova, Reggio Emilia
- Centre Hospitalier, Luxembourg, Luxembourg
- Champalimaud Foundation, Lisbon, Portugal
- Spain (15):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital del Mar, Barcelona
  - Dr Rosell Oncology Institute, Quirón Dexeus University Hospital, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castellon
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Universitari Arnau de Vilanova, Lleida
  - MD Anderson Cancer Center, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Centro Integral Oncológico Clara Campa, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Ryhov County Hospital, Jönköping
- Switzerland (4):
  - Kantonsspital Baden, Baden
  - Inselspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
  - Luzerner Kantonsspital, Division of Medical Oncology, Lucerne
- United Kingdom (11):
  - Queen Elizabeth Hospital - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Velindre NHS Trust, Cardiff
  - NHS Tayside, Ninewells Hospital, Dundee
  - Edinburgh Cancer Centre - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospital NHS Trust, Nottingham
  - Singleton Hospital - ABM University Health Board, Swansea
  - Royal Cornwall Hospital - Royal Cornwall Hospitals NHS Trust, Truro
  - Yeovil District Hospital NHS Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: sponsor's website — http://www.bigagainstbreastcancer.org